CLINICAL TRIAL: NCT03944876
Title: Botulinum Toxin Type A Blockade of the Sphenopalatine Ganglion in Treatment-refractory Chronic Cluster Headache
Acronym: BASIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); University College, London (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Catholic University of Valencia (Other); PRAXISKLINIK ULMENHOF (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/1821; 2018-003148-21 (EudraCT Number)
Record Dates: First submitted 2019-04-26; First posted 2019-05-10 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Cluster Headache
Keywords: Botulinum Toxin Type A; Sphenopalatine Ganglion Block; Autonomic Nerve Block; Injections
MeSH Terms: conditions — Cluster Headache | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox injections towards SPG (Experimental): Botulinum Toxin type A injections
  Interventions: Drug: Botulinum toxin type A
- Controls (Placebo Comparator): placebo injections
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin 25 Allergan units in 0.5 ml Sodium Chloride (NaCl) 0.9 % Braun. One injection in the headache side of the face, targeted at the sphenopalatine ganglion (SPG)
  Other Names: botox
  Arms: Botox injections towards SPG
Drug: placebo — 0.5 ml Sodium Chloride (NaCl) 0.9% Braun. One injection in the headache side of the face, targeted at the sphenopalatine ganglion (SPG)
  Other Names: Sodium Chloride
  Arms: Controls

SUMMARY:
Cluster headache is a primary headache condition characterized by clusters of one-sided, high-intensity pain attacks. The headache may be episodic or chronic. Treatment options are limited and their effects unsatisfactory. An important nerve pathway involved in the pain attacks has a switching station at the sphenopalatine ganglion (SPG) located in the depth of the facial bones. SPG is a known therapy target for cluster headache. The area can be identified on CT images, but is difficult to access due to its location. Thus, the Multiguide navigation system has been developed to enable precise delivery of the drugs that target SPG activity. In Trondheim, two phase 1 / Phase 2 study have been carried out using botulinum toxin A (Botox®) against SPG in patient with chronic cluster headache and chronic migraine. The results indicate that such a treatment strategy is safe and beneficial. The current study is a randomized, placebo-controlled, triple-blinded study to investigate whether precise single-injection of botulinum toxin A reduces the frequency of attacks in chronic cluster headache .

ELIGIBILITY:
Inclusion Criteria:

1. Informed and written consent.
2. Male or female, 18-85 years of age
3. Headache attacks fulfilling the International Classification of Headache Disorders (ICHD) III criteria for chronic cluster headache (CCH) 3.1.2.
4. Dominant headache laterality with ≥ 80% of cluster headache attacks on one side.
5. Subject reports an average of ≥ 4 cluster attacks/week on the side of their dominant headache laterality in the 3 months prior to inclusion and in the baseline period.
6. The condition is pharmacologically refractory defined as suboptimal effect or intolerable side effects or contraindication for verapamil or lithium or suboccipital steroid injection.
7. Subject agrees to maintain current preventive headache medication regimens (no change in type, frequency, or dose) during the whole study period.
8. Subject is able to differentiate concomitant headaches from cluster headache.
9. In case of women of childbearing potential (WOCBP) they have to be using highly effective contraception in a period of 4 weeks after injection.
10. Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

1. Subject has had a change in type, dosage or dose frequency of preventive headache medications ≥ two weeks prior to baseline/screening or 5 half-lives, whichever is longer.
2. Subject currently treated with occipital nerve stimulation, deep brain stimulation or other implantable device, that have changed parameters in the last month, or are unable to keep parameters stable throughout the study.
3. Current or previous treatment with implanted medical devices targeting the SPG
4. Subject has had a change in type, dosage or dose frequency of preventive headache medications during the baseline period, eg. prior to IMP administration.
5. Non-responder to both oxygen and triptan.
6. Participation in a clinical study of a new chemical entity or a prescription medicine within 2 months before study drug administration or 5 half-lives, whichever is longer.
7. Subject is currently participating or has participated in the last 3 months in another clinical study in which the subject has, is, or will be exposed to an investigational or non-investigational drug or device.
8. Allergy or hypersensitivity reactions to marcaine, lidocaine, xylocaine, adrenaline, any botulinum toxin or similar substances.
9. Abuse of drugs or alcohol.
10. Use of opioids for ≥10 days per month.
11. Treatment with pharmacological substances that may interact with BTA (aminoglycosids, spectinomycin, neuromuscular blockers, both depolarizing agents (such as succinylcholine) or non-depolarizing (tubocurarine derivates), lincosamides, polymyxins, quinidine, magnesium sulfate or anticholinestases.).
12. WOCBP that do not adhere to the requirements for HEC, as noted in inclusion criteria 9 and outlined in section 3.3.
13. Pregnancy or breastfeeding in the study period
14. Subject has undergone facial surgery in the area of the pterygopalatine fossa or zygomaticomaxillary buttress ipsilateral to the planned injection site that, in the opinion of the Investigator, may lead to an inability to properly conduct the procedure.
15. Facial anomaly or trauma which renders the procedure difficult.2
16. Subject currently has an active oral or dental abscess or a local infection at the site of injection based on present symptoms.
17. Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving the face that have been active or required treatment in the past 6 months.
18. Patients exhibiting a high degree of comorbidity and/or frailty associated with reduced life expectancy or high likelihood of hospitalization, at the discretion of the investigator.
19. Patients with comorbid psychiatric disorders with psychotic or other symptoms making compliance with the study protocol difficult, at the discretion of the investigator.
20. Patient with active infectious disease or infections that warrants special infection control measures, such as human immunodeficiency virus, tuberculosis, or chronic hepatitis B or C infection.
21. Patient with disorders that are known contraindication for Botox® treatment, especially neuromuscular disorders such as motorneuron disorders and myasthenic syndromes
22. Subject has had previous radiofrequency ablation, balloon compression, gamma knife, or chemical denervation (e.g. glycerol treatments) of the ipsilateral trigeminal ganglion or any branch of the trigeminal nerve.
23. Subject has had previous radiofrequency ablation (including non-lesional pulsed radiofrequency), balloon compression, gamma knife, or chemical denervation (e.g. glycerol treatments) of the ipsilateral SPG.
24. Subject has had blocks of short-acting anaesthetics of the ipsilateral SPG in the last 3 months.
25. Subject has undergone onabotulinumtoxinA injections of the head and/or neck in the last 3 months.
26. Subject is anticipated to require any excluded medication, device, or procedure during the study.
27. Subject has a history of bleeding disorders and in the opinion of the Investigator, may lead to an inability to properly conduct the procedure.
28. Subject has a history of coagulopathy.
29. Subject is unable to stop antithrombotic medication, eg. anticoagulants and/or antiplatelet therapy, before procedure.
30. The subject has been diagnosed with another trigeminal autonomic cephalalgia or trigeminal neuralgia.
31. The patient cannot participate or successfully complete the study, in the opinion of their healthcare provider or the investigator, for any of the following reasons:

    * mentally or legally incapacitated or unable to give consent for any reason.
    * in custody due to an administrative or a legal decision, under tutelage, or being admitted to a sanatorium or social institution.
32. The patient is a study centre employee who is directly involved in the study or the relative of such an employee.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Difference in change from baseline week 5-8 in mean number of cluster headache attacks per week at weeks 5-8 post-intervention in the treatment group versus the placebo group | week 5 through week 8 in the post-injection period
  Change from baseline to weeks 5-8 post-intervention in number of cluster headache attacks per week in the active group versus the placebo group. The number of cluster headache attacks is collected in a headache diary.

SECONDARY OUTCOMES:
Difference in occurrence of adverse events (AEs) and serious adverse events (SAEs) in the active group versus the placebo group | week 1 through week 12 in the post-injection period
  All adverse events and serious adverse events occurring in the 3 months follow up are registered in an electronic case report form (CRF). Frequency of AE and SAE are compared between the placebo group and the treatment group
Difference in change from baseline week 5-8 in mean number of cluster headache attacks per week during weeks 9-12 post-intervention in the active group versus the placebo group | week 9 through week 12 in the post-injection period
  Change from baseline to weeks 9-12 post-intervention in number of cluster headache attacks per week in the active group versus the placebo group. The number of cluster headache attacks is collected in a headache diary
Difference in change from baseline week 5-8 in mean number of cluster headache attacks per week at weeks 5-8 post-intervention in the active group versus the placebo group, in the prespecified subgroups | week 5 through week 8 in the post-injection period
  Change from baseline to weeks 5 - 8 post-intervention in number of cluster headache attacks per week comparing high versus low attack frequency and low versus high attack frequency variation in the entire baseline period. Comparisons are done between the active and the placebo group. The number of cluster headache attacks is collected in a headache diary
Difference in change from baseline week 5-8 in mean number of cluster headache attacks per week during weeks 9-12 post-intervention in the active group versus the placebo group, in the prespecified subgroups | week 9 through week 12 in the post-injection period
  Change from baseline to weeks 9-12 post-intervention in number of cluster headache attacks per week comparing high versus low attack frequency and high versus low attack frequency variation in the entire baseline period. Comparisons are done between the active and the placebo group. The number of cluster headache attacks is collected in a headache diary
Difference in the number of therapeutic responders in the active group versus the placebo group. | week 5 through week 8 in the post-injection period
  Number of therapeutic responders as defined as a ≥ 30% reduction in attack frequency, intensity or both during weeks 5 - 8 post-intervention compared to baseline week 5-8. The number in the placebo and intervention group are compared
Difference in the number of attack frequency responders | week 5 through week 8 in the post-injection period
  Number of attack frequency responders as defined as a ≥ 30% reduction in attack frequency during weeks 5-8 post-intervention compared to baseline. The number in the placebo and intervention group are compared
Difference in change from baseline week 5-8 in mean attack intensity week 5 - 8 post-intervention in the active group versus the placebo group. | week 5 through week 8 in the post-injection period
  Mean attack intensity (10-point numerical response scale - NRS) week 5-8 post intervention compared to baseline in the intervention group versus the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Geir Bråthen, md phd, Study Director — St. Olavs Hospital
Locations (5):
- Praxisklinik Ulmenhof, Hamburg, Germany
- Fondazione IRCCS Istituto Neurologico Carlo Besta (CBNI), Milan, Italy
- St Olavs Hospital, Trondheim, Norway
- Department of Neurology, University Clinic Hospital. Catholic University of Valencia, Valencia, Spain
- National Hospital of Neurology and Neurosurgery, University College of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared within 6 months after study results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after study results publication
Access Criteria: erling.tronvik@ntnu.no